CLINICAL TRIAL: NCT01786993
Title: MultiPoint Pacing IDE Study
Acronym: MPP IDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60029161/D
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-point pacing arm (Experimental): MultiPoint Pacing
  Interventions: Device: MultiPoint Pacing
- Biventricular arm (Active Comparator): Traditional Biventricular Pacing
  Interventions: Device: Traditional Biventricular Pacing

INTERVENTIONS:
Device: MultiPoint Pacing — Subjects are programmed to MPP between 3 and 9 months. MPP programming is stipulated by the Echocardiographic measurements (e.g. EA VTI) during an acute hemodynamic assessment at the 3-month visit in the MPP IDE study.
  Arms: Multi-point pacing arm
Device: Traditional Biventricular Pacing — Subjects are programmed to Quadripolar BiV pacing between 3 and 9 months using any of the 10 vectors available.
  Arms: Biventricular arm

SUMMARY:
This IDE study is a prospective, randomized, double-blind, multi-center clinical study to evaluate the safety and efficacy of patient treatment with MPP compared to patient treatment with standard BiV pacing at 9 months.

The study will be conducted at a maximum of 50 investigational centers located in the United States. A maximum of 506 subjects implanted with the Quadripolar cardiac resynchronization therapy device (CRT-D) system will be enrolled in the study.

DETAILED DESCRIPTION:
All subjects will undergo a 2 dimensional Echocardiogram within the 30 days prior to implant, and again at 3, 6 and 9 months post implant. At implant, the final LV pacing configuration is programmed using any one of the 10 available pacing vectors. The paced/sensed atrioventricular (AV) and interventricular (VV) delays may be optimized as per the site's standard of care. Subjects will continue to receive BiV therapy until the 3-month follow-up visit.

At the 3-month visit, responder status between Enrollment and 3 months will be assessed using the Clinical Composite Score (CCS). All subjects that are "Improved" using the definition outlined in the CCS will be grouped together as Responders. All subjects that are "Worsened" or "Unchanged" using the definitions outlined in the CCS will be considered as Non-responders. All subjects will undergo acute measurement of cardiac performance (e.g., Echocardiography) at various MPP combinations compared to BiV pacing. Only subjects with "equal or better" echocardiographic measurements (i.e., EA VTI measurements) with MPP feature on compared to BiV pacing will be randomized in a 1:1 ratio to one of the two arms - BiV arm or MPP arm.

At the 9-month visit, responder status will be evaluated once again using the CCS and compared to the status at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets current clinical indication for implantation of a cardiac resynchronization therapy system for treatment of heart failure or life-threatening ventricular tachyarrhythmia(s)
* Receiving a new CRT implant or undergoing an upgrade from an existing ICD or pacemaker implant with no prior LV lead placement
* Have the ability to provide informed consent for study participation and are willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Have had a recent Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) within 3 months of enrollment
* Have an existing Class I recalled lead
* Have a hypersensitivity to a single 1.0mg dose of dexamethasone sodium phosphate
* Have a classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 9 months
* Have permanent atrial fibrillation (AF)
* Have undergone a cardiac transplantation within 40 days of enrollment
* Have had a recent myocardial infarction, unstable angina within 40 days or cardiac revascularization within 3 months of implant.
* Are currently participating in a clinical investigation that includes an active treatment arm
* Are pregnant or planning to become pregnant during the duration of the study
* Have a life expectancy of less than 9 months due to any condition
* Are less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gery Tomassoni, MD, Principal Investigator — Central Baptist Hospital
Locations (49):
- United States (49):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Banner Heart Hospital, Mesa, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - Premier Cardiology, Inc, Newport Beach, California
  - Regional Cardiology Associates, Sacramento, California
  - Sutter Memorial Hospital, Sacramento, California
  - Colorado Heart & Vascular, P.C., Lakewood, Colorado
  - Cardiology Associates of Fairfield County, PC, Norwalk, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Bay Area Cardiology Associates PA, Brandon, Florida
  - Watson Clinic Center, Lakeland, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St. Joseph's Hospital, Atlanta, Georgia
  - HeartCare Midwest, Peoria, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Thoracic Cardio Healthcare Foundation, Lansing, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Novant Health Heart and Vascular Research Institute, Charlotte, North Carolina
  - Wake Forest University Medical Center Clinical Sciences, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Cardiology Center of Amarillo, L.L.P, Amarillo, Texas
  - Austin Heart, Austin, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Cardiovascular Associates, LTD, Virginia Beach, Virginia
  - Aurora Medical Group, Milwaukee, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The study results will be presented at HRS Late-Breaking Clincial Trials Session in May, 2016

REFERENCES:
- [Derived] Varma N, Baker J 2nd, Tomassoni G, Love CJ, Martin D, Sheppard R, Niazi I, Cranke G, Lee K, Corbisiero R. Left Ventricular Enlargement, Cardiac Resynchronization Therapy Efficacy, and Impact of MultiPoint Pacing. Circ Arrhythm Electrophysiol. 2020 Nov;13(11):e008680. doi: 10.1161/CIRCEP.120.008680. Epub 2020 Oct 7. PMID 33028082
- [Derived] Niazi I, Baker J 2nd, Corbisiero R, Love C, Martin D, Sheppard R, Worley SJ, Varma N, Lee K, Tomassoni G; MPP Investigators. Safety and Efficacy of Multipoint Pacing in Cardiac Resynchronization Therapy: The MultiPoint Pacing Trial. JACC Clin Electrophysiol. 2017 Dec 26;3(13):1510-1518. doi: 10.1016/j.jacep.2017.06.022. Epub 2017 Sep 27. PMID 29759832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 506 subjects at 49 investigational centers located in the U.S. A patient was considered enrolled upon signing informed consent. The first subject was enrolled on April 25, 2013. The study was double-blinded (the study subjects and the authorized personnel conducting the NYHA Class and Patient Global assessments were blinded).
Pre-assignment Details: 455 out of 469 subjects with an attempted implant (97% success rate) received Quadripolar BiV pacing between implant and 3 months. At 3 months, responder status was assessed per Clincial Composite Score and 1:1 randomziation was stratified by responder status. 381 patients were randomized to either BiV (n = 180) or MPP (n = 201) at 3 months.
Groups:
- Multi-point Pacing Arm: Subjects were programmed to MPP between 3 and 9 months. MPP programming was stipulated by the Echocardiographic measurements (e.g. EA VTI) during an acute hemodynamic assessment at the 3-month visit in the MPP IDE study.
- Biventricular Arm: Subjects were programmed to Quadripolar BiV pacing between 3 and 9 months using any of the 10 vectors available.
Period: Overall Study
Arm/Group | Multi-point Pacing Arm | Biventricular Arm
Started | 201 | 180
Per Protocol Population at 9 Months | 189 | 170
Completed | 189 | 170
Not Completed | 12 | 10
Not completed — Death | 6 | 7
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject Non-Compliance | 1 | 0
Not completed — System Explant | 1 | 0
Not completed — Hospice Admission | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 381 subjects were randomized at 3 months, of whom 180 were in the BiV arm and 201 were in the MPP arm.
Groups:
- MultiPoint Pacing Arm: Subjects were programmed to MPP between 3 and 9 months. MPP programming was stipulated by the Echocardiographic measurements (e.g. EA VTI) during an acute hemodynamic assessment at the 3-month visit in the MPP IDE study.
- Total: Total of all reporting groups
Arm/Group | MultiPoint Pacing Arm | Biventricular Arm | Total
Number analyzed (Participants) | 201 | 180 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10) | 68 (10) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 61 | 134
  Male | 128 | 119 | 247
Region of Enrollment [Number; unit: participants]
  United States | 201 | 180 | 381
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 10 | 5 | 15
  Non-Hispanic or Latino | 191 | 175 | 366
RACE [Number; unit: participants]
  White | 176 | 163 | 339
  Black or African American | 19 | 16 | 35
  Asian | 2 | 0 | 2
  Other | 4 | 1 | 5
QRS Duration [Mean (Standard Deviation); unit: ms] | 158 (24) | 154 (20) | 156 (22)
QRS Morphology [Number; unit: participants]
  Left Bundle Branch Block (LBBB) | 146 | 139 | 285
  Right Bundle Branch Block (RBBB) | 21 | 20 | 41
  Interventricular Conduction Delay (IVCD) | 32 | 21 | 53
  Unknown | 2 | 0 | 2
Cardiomyopathy Etiology [Number; unit: participants]
  Ischemic | 96 | 88 | 184
  Non-ischemic | 103 | 91 | 194
  None | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Freedom From System-related Complications Through 9 Months Compared to an Objective Performance Criterion
Description: A system related complication is a complication related to the Quadripolar CRT-D device system which includes pulse generator and leads, as adjudicated by an independent Clinical Events Committee (CEC). All subjects who had an attempted implant or a successful Quadripolar system implant were included in the analysis of this safety endpoint.
Time Frame: Implant to 9 months
Population: Of 469 subjects who underwent an attempted implant, 31 subjects experienced a system-related complication between implant and 9 months (13 were LV lead-related, 16 were RA/RV lead-related and 3 were Quadripolar CRT-D pulse generator related. One subject experienced more than one category of complication).
Measure: Number (95% Confidence Interval); unit: Event-Free Probability
Groups:
- BiV/MPP Patients: Of 469 subjects who underwent an attempted implant, 31 subjects experienced a system-related complication between implant and 9 months (13 were LV lead-related, 16 were RA/RV lead-related and 3 were Quadripolar CRT-D pulse generator related. One subject experienced more than one category of complication).
Arm/Group | BiV/MPP Patients
Number analyzed (Participants) | 469
Event-Free Probability | 0.932 [0.904 to 0.951]
Statistical Analysis 1: Comparison: BiV/MPP Patients; The hypothesis is formally expressed as: H0: Freedom from system-related complications through 9 months ≤ 75% Ha: Freedom from system-related complications through 9 months > 75%; Test type: Superiority or Other; Event-Free Probability = 0.932, 95% CI 2-sided [0.904 to 0.951]

2. Primary Outcome: Percentage of Non-responders With MPP Compared to Biventricular Pacing
Description: The hypothesis is that the non-response rate to CRT therapy in the MPP therapy arm is not inferior to the non-response rate in the BiV arm between 3 and 9 months post-implant. Responder status was assessed using the Clinical Composite Score (CCS). A patient's CCS was classified as worsened, improved or unchanged based on the definitions below:
  * Worsened - patient died due to cardiovascular reasons, experienced a HF event, demonstrated worsening in NYHA class, or had worsening of PGA score compared to the last observation
  * Improved - patient survived without a HF event, and demonstrated either improvement in NYHA class or improvement in PGA score, or both compared to the last observation.
  * Unchanged - patient was neither improved nor worsened
  For patients who were responders at the 3-month visit, those who were "Improved" and "Unchanged" between 3 and 9 months were classified as responders, whereas those who were "Worsened" were grouped together as non-responders.
Time Frame: 3 months to 9 months
Measure: Number; unit: percentage of patients
Groups:
- MultiPoint Pacing Arm: MultiPoint Pacing
  MultiPoint Pacing: Subjects are programmed to MPP between 3 and 9 months. MPP programming is stipulated by the Echocardiographic measurements (e.g. EA VTI) during an acute hemodynamic assessment at the 3-month visit in the MPP IDE study.
Arm/Group | MultiPoint Pacing Arm | Biventricular Arm
Number analyzed (Participants) | 201 | 180
percentage of patients | 29.9 | 25
Statistical Analysis 1: Comparison: MultiPoint Pacing Arm vs Biventricular Arm; H0: (Non-responder rate in the BiV arm between 3 M randomization and 9 M) - (Non-responder rate in the MPP arm between 3 M randomization and 9 M) ≤ -0.15 Ha: (Non-responder rate in the BiV arm between 3 M randomization and 9 M) - (Non-responder rate in the MPP arm between 3 M randomization and 9 M) > -0.15 The null hypothesis will be rejected at the 2.5% significance level if the lower one-sided 97.5% confidence bound for the difference in the proportions is above -0.15; Test type: Non-Inferiority or Equivalence — Assuming a binomial distribution with a 44% probability for non-responders between 3 months and 9 months in both study arms, the sample size required for 85% power to reject the null hypothesis at the 5% significance level is 394. To adjust for a potential net crossover of 15% and an overall attrition rate of 20%, the total number of patients required to be enrolled in this study is 506; p = 0.0131, normal approximation for binomial dist; Difference of proportions = -0.049, 97.5% CI 1-sided [lower limit -0.138]

ADVERSE EVENTS:
Time Frame: 3-month randomization to 9 months
Description: * Serious Adverse Events: Events that require invasive intervention (e.g. lead dislodgment requiring repositioning).
  * Other Adverse Events: Events that can be managed without invasive intervention (e.g., oversensing or loss of pacing capture, which is remedied by reprogramming of the pulse generator).
Arm/Group | MultiPoint Pacing Arm | Biventricular Arm
Serious Adverse Events (participants affected / at risk) | 4/201 | 3/180
Other Adverse Events (participants affected / at risk) | 40/201 | 5/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MultiPoint Pacing Arm (N=201) | Biventricular Arm (N=180)
LV Lead Dislodgement or Migration (Cardiac disorders) | 1 (1) | 3 (3)
RA/RV Lead Dislodgement or Migration (Cardiac disorders) | 1 (2) | 0 (0)
Pulse Generator Erosion/Extrusion (Cardiac disorders) | 1 (1) | 0 (0)
Generator Malfunction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MultiPoint Pacing Arm (N=201) | Biventricular Arm (N=180)
LV Lead Elevated Pacing Thresholds (Cardiac disorders) | 3 (3) | 0 (0)
LV Lead Loss of Capture (Cardiac disorders) | 2 (2) | 0 (0)
Phrenic Nerve/Diaphragmatic Stimulation Related to LV Lead (Cardiac disorders) | 21 (25) | 0 (0)
Rise in Threshold And Exit Block Related to LV Lead (Cardiac disorders) | 1 (1) | 0 (0)
RA/RV Lead Elevated Pacing Thresholds (Cardiac disorders) | 1 (1) | 0 (0)
RA/RV Lead Loss of Capture (Cardiac disorders) | 1 (1) | 0 (0)
RA/RV Lead Oversensing (Cardiac disorders) | 1 (1) | 2 (2)
Artifact Observed on Atrial Channel (Cardiac disorders) | 10 (10) | 0 (0)
Discomfort Around Device (Cardiac disorders) | 1 (1) | 0 (0)
Intolerance to MPP Pacing (Cardiac disorders) | 1 (1) | 0 (0)
Pulse Generator Oversensing (Cardiac disorders) | 1 (1) | 2 (2)
Pacemaker Mediated Tachycardia (PMT) (Cardiac disorders) | 1 (1) | 0 (0)
Intolerance to BiV Pacing (Cardiac disorders) | 0 (0) | 1 (1)
Thrombo-Embolic Event (Cardiac disorders) | 1 (1) | 0 (0)
Erythema to Lateral Aspect of Incision Site (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less